CLINICAL TRIAL: NCT02220270
Title: A Prospective, Multi-center Study to Evaluate the Safety and Performance of the Hyperion™ ASD and PDA Closure Systems.
Brief Title: Hyperion™ International Registry Trial
Acronym: COM-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Cardiovascular Research Center (Network)
Collaborators: Comed B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: COM-01 V1.0 17 June 2014
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Septal Defects; Patent Ductus Arteriosus
MeSH Terms: conditions — Heart Septal Defects, Atrial; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with PDA or ASD
  Interventions: Device: ASD and PDA closure

INTERVENTIONS:
Device: ASD and PDA closure

SUMMARY:
The purpose of this study is to determine the safety, performance and efficacy of the Hyperion™ Occluder Systems during treatment of ASD and PDA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has ASD or PDA documented by a Transoesophagial echocardiography (TEE) or a Transthoracic echocardiography (TTE) and indication for closure that is amenable to treatment with the Hyperion™ ASD or PDA occluder
* For PDA: Patient age ≥ 1 year old
* For ASD: Patient weighting ≥15 kg of any age
* Patient is willing and able to comply with specified follow-up evaluations
* Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written Notice of Informed Consent, approved by the appropriate Ethics Committee (EC)

Exclusion Criteria:

* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test
* Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year)
* Patient has a known hypersensitivity or contraindication to aspirin, heparin, and/or contrast sensitivity that cannot be adequately pre-medicated
* Currently participating in another clinical study
* Active endocarditis, active bacterial infection, or other infection producing bacteremia or sepsis
* Congenital or structural heart disease other than ASD or PDA
* Thrombus at the intended site of implant or documented venous thrombosis in venous access
* Severe pulmonary hypertension
* Vascular anatomy unable to accommodate the appropriate-sized sheath for device introduction
* ASD or PDA anatomy non suitable for the Hyperion™ closure device
* Confinement to bed (increased risk for clot formation)
* Prior cardiac implantation of cardiac devices for ASD or PDA closure

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who comes to hospital for ASD or PDA closure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Success of implantation | 30 days
  Success of implantation without death, stroke, any device embolization, puncture site bleeding requiring surgical repair or blood transfusion and without any other device or procedure related MAE at 30 days
Device success | 6 months
  Device success defined as ASD or PDA closure at 6 months post procedure by a Transthoracic echocardiography (TTE) or a Transesophageal echocardiography (TEE).

SECONDARY OUTCOMES:
Major Adverse Events | 30 days, 6 and 12 months
  * Major Adverse Events at 6 and 12 months defined as composite rate of all death, stroke, any device embolization, puncture site bleeding requiring surgical repair or blood transfusion at discharge and any other device or procedure related MAE.
  * Components of Major Adverse Events at discharge, 30 days, 6, and 12 months.
Procedure success | 6 months
  Procedure success defined as successful deployment of the Hyperion™ Closure System in the patient's ASD and PDA, closure (residual shunt < 3mm) at 6 months.

CONTACTS AND LOCATIONS:
Locations (10):
- Algeria (3):
  - CHU Frantz-Fanon, Blida
  - Radjah Clinic, Sétif
  - Centre Médico-chirurgical infantile Bou Ismail, Tipasa
- China (2):
  - Anzhen Hospital, Beijing
  - Shanghai Children's Medical Center, Shanghai
- France (4):
  - Hôpital cardiologique Haut-Leveque (CHU Bordeaux), Bordeaux
  - Hôpital Privé Jacques Cartier, Massy
  - Hopital Necker Enfants Malades, Paris
  - American Memorial Hospital, Reims
- CardioVascular Center Frankfurt, Frankfurt, Germany